CLINICAL TRIAL: NCT06575478
Title: Evaluation of Fuling Yunhua Granules and Dihuang Baoyuan Granules in Type 2 Diabetes Patients With Poor Blood Glucose Control After Diet and Exercise Intervention: a Multi-center, Randomized, Double-blind, Placebo-controlled Clinical Study
Brief Title: Evaluation of Fuling Yunhua Granules and Dihuang Baoyuan Granules in Drug Naive Type 2 Diabetes Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Supreme Life Pharmaceutical Technology Co., Ltd. (Industry)
Collaborators: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JYHS-BAIIT-Pro-24001
Record Dates: First submitted 2024-08-19; First posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2; Diabetes; Type2diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- prescription ABA (Experimental): Fuling Yunhua Granules and Dihuang Baoyuan Granules
  Interventions: Drug: Fuling Yunhua Granules
- prescription ABA-matched placebo (Placebo Comparator): Fuling Yunhua Granules placebo and Dihuang Baoyuan Granules placebo
  Interventions: Drug: Fuling Yunhua Granules matched placebo
- prescription BAB (Experimental): Fuling Yunhua Granules and Dihuang Baoyuan Granules
  Interventions: Drug: Dihuang Baoyuan Granules
- prescription BAB-matched placebo (Placebo Comparator): Fuling Yunhua Granules placebo and Dihuang Baoyuan Granules placebo
  Interventions: Drug: Dihuang Baoyuan Granules matched placebo

INTERVENTIONS:
Drug: Fuling Yunhua Granules — Fuling Yunhua Granules
  Other Names: prescription A
  Arms: prescription ABA
Drug: Fuling Yunhua Granules matched placebo — Fuling Yunhua Granules placebo
  Other Names: prescription A matched placebo
  Arms: prescription ABA-matched placebo
Drug: Dihuang Baoyuan Granules — Dihuang Baoyuan Granules
  Other Names: prescription B
  Arms: prescription BAB
Drug: Dihuang Baoyuan Granules matched placebo — Dihuang Baoyuan Granules placebo
  Other Names: prescription B matched placebo
  Arms: prescription BAB-matched placebo

SUMMARY:
The goal of this investigator-initiated clinical trial is to investigate the efficacy and safety of sequential therapy of Fuling Yunhua Granules (prescription A) and Dihuang Baoyuan Granule (prescription B) in the treatment of type 2 diabetes patients with poor glycemic control after diet and exercise intervention.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study, including a up to 2-week screening period, a 1-week baseline period, a 12-week treatment period and a 1-week follow-up period.

72 participants who meet the enrollment requirements will enter the baseline period, during which 7 days of CGM data will be collected. After entering the treatment period, participants will be randomly assigned to prescription ABA group, prescription ABA-matched placebo group, prescription BAB group and prescription BAB-matched placebo group in a ratio of 2:1:2:1 and receive corresponding treatment.

It is expected that an interim analysis will be conducted after 30 participants have completed 4 weeks of treatment and 4 weeks of their data is obtained. Based on the CGM data of the participants in the 4th week of treatment, the change of TIR in the 4th week compared with the baseline will be analyzed, and the IDMC will make a decision based on the results of this analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years (inclusive), male or female;
2. Patients diagnosed with T2DM ≥ 8 weeks according to the 2020 WHO diagnostic criteria and classification;
3. Have controlled blood sugar through diet and exercise for 3 months before screening and did not receive any hypoglycemic drugs, or used hypoglycemic drugs for no more than 2 weeks within 3 months before screening and did not use hypoglycemic drugs within 1 month before screening;
4. Body mass index (BMI) ≥ 19 kg/m2;
5. Glycated hemoglobin (HbA1c) ≥ 7.0% and < 10.5% at screening;
6. Fasting plasma glucose (FPG) < 13.9 mmol/L at screening;
7. Able to understand the procedures and methods of this study, willing to strictly abide by the clinical research protocol to complete this study, and voluntarily sign the ICF

Exclusion Criteria:

1. Non-type 2 diabetes: type 1 diabetes, gestational diabetes, special types of diabetes;
2. History of acute complications of diabetes within 6 months before screening (diabetic ketoacidosis, diabetic hyperglycemic hyperosmolar syndrome or lactic acidosis, etc.);
3. History of chronic complications of diabetes with unstable condition or requiring treatment within 6 months before screening (proliferative retinal disease, severe diabetic neuropathy or intermittent claudication, etc.);
4. Experienced more than 3 episodes of grade 3 hypoglycemia within 6 months before screening;
5. Have used systemic (intravenous, oral or intra-articular) glucocorticoids continuously or cumulatively for ≥ 7 days within 3 months before screening;
6. Severe infection within 3 months before screening;
7. Diagnosed with malignant tumors within 5 years before screening (except for cured basal cell carcinoma of the skin or carcinoma in situ of the cervix);
8. Severe cardiovascular disease, such as heart failure (New York Heart Association [NYHA] grade III-IV), myocardial infarction, coronary artery bypass grafting or percutaneous coronary intervention, occurred within 6 months before screening, Sustained and clinically significant arrhythmia (such as second- or third-degree atrioventricular block or QTc interval prolongation ≥470 ms in men and ≥480 ms in women), acute coronary syndrome or transient ischemic attack or stroke wait;
9. Suffering from diseases that may significantly affect drug absorption, distribution, metabolism and excretion within 6 months before screening: inflammatory bowel disease, peptic ulcer, history of gastrointestinal or rectal bleeding, history of important gastrointestinal surgery (such as : Gastrectomy, gastrointestinal anastomosis, or intestinal resection), etc.;
10. Accompanied by thyroid dysfunction that cannot be controlled with stable drug dosage during screening;
11. History of hypertension and take antihypertensive treatment regularly for more than 4 weeks but still have poor blood pressure control, with systolic blood pressure >160 mmHg and/or diastolic blood pressure >100 mmHg;
12. History of organ transplantation or severe autoimmune diseases in the past or present;
13. History of clinically significant drug allergy or atopic allergic disease (asthma, urticaria, eczematous dermatitis);
14. History of major surgery (intrathoracic, intracranial, abdominal, etc.) within 6 months before screening, or those who plan to undergo surgery during the study that may affect study completion or compliance;
15. Any laboratory test meets any of the following criteria during screening:

    Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > upper limit of normal (ULN) × 2.5 times Glomerular filtration rate (eGFR) calculated using the CKD-EPI formula < 60 mL/min /1.73m2 Total bilirubin (TBIL)>ULN×1.5 times Fasting triglyceride (TG)>5.7 mmol/L Fasting C-peptide <0.8 ng/ml (or 0.26 nmol/L)
16. Those who are positive for hepatitis B surface antigen during screening (except those whose quantitative test results of hepatitis B virus deoxyribonucleic acid [HBV-DNA] are lower than the lower limit of the detection reference range and who are not using anti-hepatitis B virus drugs during screening), or who are receiving anti-hepatitis B virus drug treatment , or those who are hepatitis C virus (HCV) antibody positive, or human immunodeficiency virus (HIV) antibody positive, or Treponema pallidum antibody positive;
17. Blood donation or massive blood loss (>400 mL) within 3 months before screening;
18. Pregnant or lactating women, or men or women of childbearing potential who plan to become pregnant during the study or are unwilling to take medically recognized contraceptive measures;
19. History of alcohol, tobacco addiction or drug abuse is known or suspected at the time of screening;
20. Participated in any interventional drug clinical research within 3 months before screening;
21. Allergic to study drugs and their ingredients;
22. Participants who the researcher believes have any other factors that are inappropriate for participating in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c concentrations (%) from baseline | 12 weeks
  Change in HbA1c concentrations (%) from baseline

SECONDARY OUTCOMES:
Change in FPG (mmol/L) from baseline | 12 weeks
  Change in FPG (mmol/L) from baseline
The proportion of participants who achieved HbA1c target | 12 weeks
  The proportion of participants who achieved HbA1c target (HbA1c<7.0% and <6.5% Patient percentage)
Changes in TIR from baseline | 7 days
  Changes in TIR from baseline
Changes in TBR from baseline | 7 days
  Changes in TBR from baseline
Changes in TAR from baseline | 7 days
  Changes in TAR from baseline
Changes in MAGE from baseline | 7 days
  Changes in MAGE from baseline
Changes in fasting lipid profiles | 12 weeks
  Changes in fasting lipid profiles from baseline(mmol/L)
Change in weight | 12 weeks
  Change in weight from baseline(kg)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.